CLINICAL TRIAL: NCT03033420
Title: Reducing the Rate and Duration of Re-ADMISsions Among Patients With Unipolar Disorder and Bipolar Disorder Using Smartphone-based Monitoring and Treatment - The RADMIS Trials
Acronym: RADMIS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Psychiatric Centre Rigshospitalet (Other)
Collaborators: Technical University of Denmark (Other)
Responsible Party: Principal Investigator, Maria Faurholt-Jepsen, Medical Doctor, Psychiatric Centre Rigshospitalet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RADMIS
Record Dates: First submitted 2017-01-13; First posted 2017-01-26 (Estimated); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Affective Disorders; Unipolar Depression; Bipolar Disorder
Keywords: Unipolar disorder; Bipolar disorder; Randomized controlled trial; Smartphone; Re-admission; CBT
MeSH Terms: conditions — Mood Disorders; Depressive Disorder; Bipolar Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): A smartphone-based monitoring system including a) an integrated feedback loop between patients and clinicians and b) context-aware CBT modules
  Interventions: Device: A smartphone-based monitoring system including a) an integrated feedback loop between patients and clinicians and b) context-aware CBT modules
- Control group (No Intervention): Treatment-as-usual

INTERVENTIONS:
Device: A smartphone-based monitoring system including a) an integrated feedback loop between patients and clinicians and b) context-aware CBT modules — A smartphone-based monitoring system including a) an integrated feedback loop between patients and clinicians and b) context-aware CBT modules
  Other Names: Monsenso
  Arms: Intervention group

SUMMARY:
Unipolar and bipolar disorder combined account for nearly half of all morbidity and mortality due to mental and substance use disorders, and burden society with the highest health care costs of all psychiatric and neurological disorders. Among these, costs due to psychiatric hospitalization is a major burden. Smartphones comprise an innovative and unique platform for monitoring and treatment of depression and mania.

The RADMIS trials use a randomized controlled single-blind parallel-group design. Patients with unipolar or bipolar disorder discharged from psychiatric hospitals in The Capital Region of Denmark are invited to participate. Patients are at discharge from the psychiatric hospitals randomized, separately according to psychiatric diagnosis (thus, the RADMIS trial consists of two separate trials according to diagnosis, bipolar disorder or unipolar disorder), to: 1) a smartphone-based monitoring system including a) an integrated feedback loop between patients and clinicians and b) context-aware CBT modules (intervention group) or 2) treatment-as-usual (control group) for a 6-months trial period. The trial is started in March 2017. The outcomes are 1) differences in the number and duration of re-admissions between the intervention group and the control group (primary), 2) differences in severity of depressive and manic symptoms (manic symptoms only for patients with bipolar disorder); differences in psychosocial functioning; and differences in number of affective episodes between the intervention group and the control group (secondary), and 3) differences in perceived stress, quality of life, self-rated depressive symptoms, self-rated manic symptoms (only for patients with bipolar disorder), recovery, empowerment, adherence to medication, well-being, ruminations, worrying, and satisfaction between the intervention group and the control group (tertiary).

DETAILED DESCRIPTION:
Background Unipolar and bipolar disorder combined account for nearly half of all morbidity and mortality due to mental and substance use disorders, and burden society with the highest health care costs of all psychiatric and neurological disorders. Among these, costs due to psychiatric hospitalization are a major burden. Smartphones comprise an innovative and unique platform for monitoring and treatment of depression and mania. No prior trial has investigated whether the use of a smartphone-based system can prevent re-admission among patients discharged from hospital.

Methods The RADMIS trials use a randomized controlled single-blind parallel-group design. Patients with unipolar disorder and patients with bipolar disorder are invited to participate in each their trial when discharged from psychiatric hospitals in The Capital Region of Denmark following an affective episode and randomized to either 1) a smartphone-based monitoring system including a) an integrated feedback loop between patients and clinicians and b) context-aware CBT modules (intervention group) or 2) standard treatment (control group) for a 6-months trial period. The trial is started in March 2017. The outcomes are 1) differences in the number and duration of re-admissions between the intervention group and the control group (primary), 2) differences in severity of depressive and manic symptoms (manic symptoms only for patients with bipolar disorder); differences in psychosocial functioning; and differences in number of affective episodes between the intervention group and the control group (secondary), and 3) differences in perceived stress, quality of life, self-rated depressive symptoms, self-rated manic symptoms (only for patients with bipolar disorder), recovery, empowerment, adherence to medication, well-being, ruminations, worrying, and satisfaction between the intervention group and the control group (tertiary).

Analysis Recruitment is ongoing.

Discussion If the smartphone-based monitoring system is proved effective in reducing the rate and duration of re-admissions there will be basis for using a system of this kind in the treatment of unipolar and bipolar disorder in general and in a larger scale.

ELIGIBILITY:
Inclusion Criteria:

* Unipolar disorder or bipolar disorder diagnoses according to ICD-10
* Patients who are discharged from a psychiatric hospital in The Capital Region of Denmark following an affective episode (depression or mania)

Exclusion Criteria:

* Pregnancy
* A lack of Danish language skills

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2017-05-15 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Number of re-admissions | 6 months trial period
  Differences in the number of re-admissions between the intervention group and the control group. Data will be collected from Danish registers.
Duration of re-admissions | 6 months trial period
  Differences in the duration of re-admissions between the intervention group and the control group.

SECONDARY OUTCOMES:
Severity of depressive symptoms | 6 months trial period
  Differences in the severity of depressive (The Hamilton Depression Rating Scale) symptoms between the intervention group and the control group.
Severity of manic symptoms | 6 months trial period
  Differences in the severity of manic (The Young Mania Rating Scale) symptoms between the intervention group and the control group.
Psychosocial functioning | 6 months trial period
  Differences in psychosocial functioning (The Psychosocial Functioning Assessment Short Test - FAST) between the intervention group and the control group.
Number of affective episodes | 6 months trial period
  Differences in the number of affective episodes between the intervention group and the control group.

OTHER OUTCOMES:
Perceived stress | 6 months trial period
  Differences in perceived stress (The Cohen's Perceived stress scale) between the intervention group and the control group.
Quality of life | 6 months trial period
  Differences in quality of life (The WHO Quality of Life-BREF) between the intervention group and the control group.
Self-rated manic symptoms | 6 months trial period
  Differences in self-rated manic symptoms (The Altman Self Rating scale for Mania) between the intervention group and the control group.
Self-rated depressive symptoms | 6 months trial period
  Differences in self-rated depressive symptoms (The Becks Depressive Inventory) between the intervention group and the control group.
Self-rated depressive symptoms | 6 months trial period
  Differences in self-rated depressive symptoms (The Hamilton Depression Self-rating Scale 6-item) between the intervention group and the control group.
Recovery | 6 months trial period
  Differences in recovery (The Recovery Assessment Scale) between the intervention group and the control group.
Empowerment | 6 months trial period
  Differences in empowerment (Rogers empowerment scale) between the intervention group and the control group.
Adherence to medication | 6 months trial period
  Differences in adherence to medication (The Medicine Adherence Rating Scale) between the intervention group and the control group.
Well-being | 6 months trial period
  Differences in well-being according (The WHO (five) well-being index) between the intervention group and the control group.
Rumination | 6 months trial period
  Differences in rumination (The Rumination Response Scale) between the intervention group and the control group.
Worrying | 6 months trial period
  Differences in worrying (The Penn State Worry Questionnaire) between the intervention group and the control group.
Satisfaction | 6 months trial period
  Differences in satisfaction (The Verona Satisfaction Scale-Affective Disorder) between the intervention group and the control group.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Faurholt-Jepsen, MD, Principal Investigator — Psychiatric Center Copenhagen, Denmark
Locations (1):
- Psychiatric Center Copenhagen, Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Faurholt-Jepsen M, Busk J, Tonning ML, Rohani D, Bardram JE, Kessing LV. Mood, Activity, and Instability in Bipolar Disorder and Unipolar Disorder-An Exploratory Post Hoc Study Using Digital Data. Acta Psychiatr Scand. 2025 Mar;151(3):426-433. doi: 10.1111/acps.13771. Epub 2024 Dec 1. PMID 39617464
- [Derived] Faurholt-Jepsen M, Frost M, Martiny K, Tuxen N, Rosenberg N, Busk J, Winther O, Bardram JE, Kessing LV. Reducing the rate and duration of Re-ADMISsions among patients with unipolar disorder and bipolar disorder using smartphone-based monitoring and treatment - the RADMIS trials: study protocol for two randomized controlled trials. Trials. 2017 Jun 15;18(1):277. doi: 10.1186/s13063-017-2015-3. PMID 28619114